CLINICAL TRIAL: NCT01840202
Title: Correlation Between Submacular and Peripapillary Choroidal Tissue and Ocular Blood Flow in Glaucoma Patients
Brief Title: Ocular Blood Flow in Glaucoma Patients - the Leuven Eye Study
Status: Completed | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: S140213
Record Dates: First submitted 2013-04-17; First posted 2013-04-25 (Estimated); Last update posted 2015-05-29 (Estimated); Status verified 2013-01

CONDITIONS: Open Angle Glaucoma; Normal Tension Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle; Low Tension Glaucoma

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Control: Healthy volunteers with no family history of glaucoma, an increased or asymmetrical cup/disc ratio or any other optic disc structural change (notching, disc hemorrhage) or an intraocular pressure (IOP) above 21 mmHg that could suggest possible glaucoma suspects.
- Primary open-angle glaucoma: Patients with a characteristic optic disc damage (based on cup/disc ratio, thinning of neuroretinal rim, notching, disk hemorrhages, etc.) and visual field defects, with at least one measurement of IOP of >21 mmHg required
- Normal Tension Glaucoma: Patients with a characteristic optic disc damage (based on cup/disc ratio, thinning of neuroretinal rim, notching, disk hemorrhages, etc.) and visual field defects, with at maximum recorded IOP of < 21 mmHg

SUMMARY:
Glaucoma is a leading cause of blindness worldwide, whose treatment - intraocular pressure lowering - is only partially effective in preventing disease progression. Accordingly, other variables, such as ocular blood flow-related factors, have been implicated in disease pathogenesis. However, most findings involving vascular variables come from partial, small-scale studies. Furthermore, recent technological advances have identified a number of ocular blood flow variables that have yet to be tested in large scale trials. Therefore, a study that specifically aims at uncovering the role of vascular aspects in glaucoma is needed.

For this purpose, a cross-sectional, observational case-control study will be conducted in the University Hospitals Leuven. This will be the largest-yet study on the subject, involving more than 750 patients. This will allow the creation of a specific cohort of patients where the vascular aspects are thought to be particularly important (low-tension glaucoma). It will use the largest combination yet of vascular-related measuring techniques (dynamic contour tonometry, optic coherent tomography, colour Doppler imaging and retinal oximetry)

DETAILED DESCRIPTION:
1. Demographic and clinical ophthalmology-related examination data will be collected, including intraocular pressure measurement using dynamic contour tonometry
2. Visual field testing will be performed.
3. Structural damage will be documented by a retinal nerve fiber layer analysis (through Heidelberg Retinal Tomograph)
4. High Definition Optical coherent tomograph imaging of the submacular and peripapillary choroidal thickness will be performed.
5. Color Doppler Imaging of the retrobulbar vessels will be performed, with analysis of the Doppler waveform (peak systolic, end diastolic velocities and resistivity index)
6. Retinal oximetry will be performed with the analysis of the arterial and venous saturations of retinal vessels

ELIGIBILITY:
Inclusion Criteria:

* individuals over 18 years old
* willing to sign an informed consent and able to comply with the requirements of the study
* having no other ocular diseases besides glaucoma

Exclusion Criteria:

* history of ocular trauma
* intraocular surgery (except for cataract surgery)
* eye disease (except glaucoma)
* systemic diseases with ocular involvement like diabetes

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Tertiary referral center
Sampling Method: Probability Sample
Enrollment: 770 (Actual)
Dates: Start 2013-02; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
Comparison of the Retrobulbar Arteries Doppler Waveform between glaucoma patients and healthy controls | Participants will be followed for the duration of hospital stay, an expected average of 2 hours

CONTACTS AND LOCATIONS:
Overall Officials: Ingeborg Stalmans, MD, PhD, Principal Investigator — UZ Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium

REFERENCES:
- [Derived] Van Keer K, Abegao Pinto L, Willekens K, Stalmans I, Vandewalle E. Correlation Between Peripapillary Choroidal Thickness and Retinal Vessel Oxygen Saturation in Young Healthy Individuals and Glaucoma Patients. Invest Ophthalmol Vis Sci. 2015 Jun;56(6):3758-62. doi: 10.1167/iovs.14-16225. PMID 26066744